CLINICAL TRIAL: NCT00984295
Title: An Open, Randomized, Multicenter Study of the Safety, Tolerability, and Immunogenicity of Frozen MMRV Given Concomitantly Versus Nonconcomitantly With Other Pediatric Vaccines in Healthy Children 12 to 15 Months of Age
Brief Title: Frozen ProQuad Administered Concomitantly Versus Nonconcomitantly With Other Pediatric Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V221-013; 2009_666
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Results first posted 2010-02-25 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Measles; Mumps; Rubella; Varicella
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox | interventions — measles, mumps, rubella, varicella vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): ProQuad + Tripedia + Comvax at Day 0 (Concomitant)
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live; Biological: Comparator: Tripedia; Biological: Comparator: Comvax
- 2 (Experimental): ProQuad at Day 0, Tripedia + Comvax at Day 42(Nonconcomitant)
  Interventions: Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live; Biological: Comparator: Tripedia; Biological: Comparator: Comvax
- 3 (Active Comparator): Varivax + M-M-R II at Day 0, Tripedia + Comvax at Day 42 (Control)
  Interventions: Biological: Comparator: Tripedia; Biological: Comparator: Comvax; Biological: Comparator: Varivax; Biological: Comparator: M-M-R II

INTERVENTIONS:
Biological: Measles, Mumps, Rubella and Varicella (Oka-Merck) Virus Vaccine Live — A single 0.5 mL subcutaneous injection at Day 0
  Other Names: ProQuad
  Arms: 1; 2
Biological: Comparator: Tripedia — A single 0.5 mL intramuscular injection (at Day 0 or Day 42)
Biological: Comparator: Comvax — A single 0.5 mL intramuscular injection (at Day 0 or Day 42)
Biological: Comparator: Varivax — A single 0.5 mL subcutaneous injection at Day 0
  Arms: 3
Biological: Comparator: M-M-R II — A single 0.5 mL subcutaneous injection at Day 0
  Arms: 3

SUMMARY:
This study will assess the safety and immunogenicity of ProQuad when administered concomitantly and nonconcomitantly with Tripedia and Comvax.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Negative clinical history of varicella, zoster, measles, mumps, rubella, diptheria, tetanus, pertussis, invasive Hib disease and hepatitis B
* Had completed either a 2-dose primary series of PedvaxHIB or COMVAX or any 3-dose primary series of a licensed Hib vaccine
* Had received 2 or 3 doses of any hepatitis B vaccine or COMVAX prior to entry into trial

Exclusion Criteria:

* Previous receipt of measles, mumps, rubella or varicella vaccine either alone or in combination
* Any immune impairment or deficiency
* Recent household, daycare or school exposure to invasive Hib disease or hepatitis B
* Exposure to measles, mumps, rubella, varicella, or zoster in the 4 weeks prior to vaccination
* Vaccination with an inactive vaccine with in the past 14 days
* Vaccination with a live vaccine within the past 30 days
* Receipt of immune globulin, blood transfusion or blood-derived product in the past 3 months
* Recent history of fever or underlying medical problems

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1913 (Actual)
Dates: Start 2000-06; Primary Completion 2001-10 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Shinefield H, Black S, Thear M, Coury D, Reisinger K, Rothstein E, Xu J, Hartzel J, Evans B, Digilio L, Schodel F, Brown ML, Kuter B; 013 Study Group for ProQuad. Safety and immunogenicity of a measles, mumps, rubella and varicella vaccine given with combined Haemophilus influenzae type b conjugate/hepatitis B vaccines and combined diphtheria-tetanus-acellular pertussis vaccines. Pediatr Infect Dis J. 2006 Apr;25(4):287-92. doi: 10.1097/01.inf.0000207857.10947.1f. PMID 16567978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 clinical sites in the United States
  Date first participant visit: 27-Jun-2000
  Date last participant visit: 23-Oct-2001
Groups:
- Concomitant Group: Concomitant Group - ProQuad™ (measles, mumps, rubella, and varicella vaccine) + TRIPEDIA™ (diphtheria and tetanus toxoids and acellular pertussis vaccine) + COMVAX™ (haemophilus b conjugate and hepatitis B vaccine) administered concomitantly at separate injection sites on Day 0.
- Nonconcomitant Group: Nonconcomitant Group - ProQuad™ (measles, mumps, rubella, and varicella vaccine) administered on Day 0 and TRIPEDIA™ (diphtheria and tetanus toxoids and acellular pertussis vaccine) and COMVAX™ (haemophilus b conjugate and hepatitis B vaccine) administered concomitantly at separate injection sites on Day 42.
- Control Group: Control Group - M-M-R™ II (measles, mumps, and rubella vaccine) and VARIVAX™ (varicella virus vaccine) administered concomitantly at separate injection sites on Day 0 and TRIPEDIA™ (diphtheria and tetanus toxoids and acellular pertussis vaccine) and COMVAX™ (haemophilus b conjugate and hepatitis B vaccine) administered concomitantly at separate injection sites on Day 42.
Period: Overall Study
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Started | 949 (2 patients were incorrectly vaccinated and are excluded from this table.) | 485 | 479
Visit 1 | 949 | 485 | 479
Visit 2 | 909 | 468 | 453
Completed | 884 | 453 | 442
Not Completed | 65 | 32 | 37
Not completed — Lost to Follow-up | 31 | 12 | 13
Not completed — Protocol Violation | 2 | 1 | 4
Not completed — Withdrawal by Subject | 18 | 9 | 12
Not completed — CAE - discontinued test vaccine | 0 | 1 | 3
Not completed — Missed one or more blood samplings | 3 | 7 | 2
Not completed — Incomplete safety follow-up | 11 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group | Total
Number analyzed (Participants) | 949 | 485 | 479 | 1913
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (0.7) | 12.3 (0.7) | 12.4 (0.7) | 12.4 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 442 | 223 | 246 | 911
  Male | 507 | 262 | 233 | 1002
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 101 | 52 | 42 | 195
  Asian/Pacific | 103 | 54 | 57 | 214
  Caucasian | 678 | 336 | 342 | 1356
  Hispanic | 38 | 26 | 20 | 84
  Native American | 3 | 0 | 1 | 4
  Other | 26 | 17 | 17 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postvaccination Measles Enzyme-Linked Immunosorbent Assay (ELISA) Antibody Titer ≥120 mIU/mL
Description: Antibody Response to Measles at 6 Weeks Postvaccination for Participants Initially Seronegative (a titer <120 mIU/mL) to Measles at Baseline
Time Frame: 6 Weeks Postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to measles at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 758 | 388 | 126
Participants | 741 | 383 | 124

2. Primary Outcome: Number of Participants With Postvaccination Mumps ELISA Antibody Titer ≥10 Ab Units/mL
Description: Antibody Response to Mumps at 6 Weeks Postvaccination for Participants Initially Seronegative (a titer <10 Ab units/mL) to Mumps at Baseline
Time Frame: 6 weeks Postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to mumps at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 811 | 415 | 145
Participants | 774 | 395 | 143

3. Primary Outcome: Number of Participants With Postvaccination Rubella ELISA Antibody Titer ≥10 IU/mL
Description: Antibody Response to Rubella at 6 Weeks Postvaccination for Participants Initially Seronegative (a titer <10 IU/mL) to Rubella at Baseline
Time Frame: 6 weeks Postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to rubella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 829 | 421 | 148
Participants | 817 | 418 | 148

4. Primary Outcome: Number of Participants With Postvaccination Varicella-Zoster Virus (VZV) Glycoprotein Enzyme-Linked Immunosorbent Assay (gpELISA) Antibody Titer ≥5 gpELISA Units/mL
Description: Antibody Response to Varicella-Zoster Virus (VZV) at 6 Weeks Postvaccination for Participants Initially Seronegative (a titer <0.6 gpELISA units/mL) to VZV at Baseline
Time Frame: 6 weeks Postvaccination
Population: The per-protocol analysis set included participants
  who had pre- and post-randomization blood samples within predefined day ranges, were seronegative to
  varicella at baseline, and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 757 | 383 | 139
Participants | 679 | 348 | 130

5. Primary Outcome: Number of Participants With Postvaccination Diphtheria Vero Cell Culture Assay Antibody Titer ≥0.1 IU/mL
Description: Antibody response to Diphtheria at 6 weeks postvaccination
Time Frame: 6 weeks Postvaccination
Population: The per-protocol analysis set included participants who had pre- and post-randomization blood samples within predefined day ranges and followed protocol procedures.
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 675 | 337 | 95
Participants | 667 | 333 | 94

6. Primary Outcome: Number of Participants With Postvaccination Tetanus Enzyme Immunoassay (EIA) Antibody Titer ≥0.1 IU/mL
Description: Antibody response to Tetanus (tetanus antitoxin were measured with an indirect, noncompetitive enzyme immunoassay (EIA)) at 6 weeks postvaccination.
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 803 | 387 | 114
Participants | 796 | 386 | 114

7. Primary Outcome: Number of Participants With ≥4-fold Rise in Pertussis Toxin (PT) EIA Antibody Titer
Description: Antibody response to Pertussis Toxin (titers of pertussis toxin antibodies were measured with an indirect, noncompetitive EIA).
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 748 | 355 | 59
Participants | 554 | 321 | 56

8. Primary Outcome: Number of Participants With ≥4-fold Rise in Pertussis Filamentous Hemagglutinin (FHA) EIA Antibody Titer
Description: Antibody response to pertussis FHA(titers of pertussis filamentous hemagglutinin antibodies were measured with an indirect, noncompetitive EIA).
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 748 | 356 | 59
Participants | 502 | 309 | 53

9. Primary Outcome: Number of Participants With Postvaccination Hepatitis B (Quantitative AUSAB™ Radioimmunoassay (RIA)) Antibody Titer ≥10 mIU/mL
Description: Antibody response to Hepatitis B (titers measured using the Quantitative AUSAB™ radioimmunoassay (RIA)).
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 825 | 396 | 122
Participants | 791 | 391 | 121

10. Primary Outcome: Number of Participants With Postvaccination Haemophilus Influenzae Type B (Hib) Radioimmunoassay (RIA) Antibody Titer ≥ 1 mcg/mL
Description: Antibody response to Haemophilus influenzae type B (Hib). (Anti-polyribosylribitol phosphate (PRP) was measured by radioimmunoassay (RIA) using radiolabeled-PRP according to a standard Farr technique and with a standard provided by the U.S. FDA.)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 822 | 398 | 124
Participants | 778 | 384 | 119

11. Primary Outcome: Antibody Response to Measles at 6 Weeks Postvaccination for Participants Initially Seronegative to Measles at Baseline - Geometric Mean Titer (GMT)
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Measles. (Titers measured using Measles ELISA.)
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to measles at baseline, and followed protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 758 | 388 | 126
mIU/mL | 3504.9 [3269.7 to 3757.2] | 3506.2 [3195.7 to 3846.9] | 2562.1 [2172.2 to 3022.0]

12. Primary Outcome: Antibody Response to Mumps at 6 Weeks Postvaccination for Participants Initially Seronegative to Mumps at Baseline - GMT
Description: Postvaccination observed GMT of antibody to mumps. (Titers measured using mumps ELISA.)
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to mumps at baseline, and followed protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA Ab units/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 811 | 415 | 145
ELISA Ab units/mL | 89.4 [83.5 to 95.7] | 84.1 [76.2 to 92.8] | 98.1 [85.7 to 112.3]

13. Primary Outcome: Antibody Response to Rubella at 6 Weeks Postvaccination for Participants Initially Seronegative to Rubella at Baseline - GMT
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Rubella. (Titers measured using Rubella ELISA.)
Time Frame: 6 weeks Postvaccination
Population: Per-protocol analysis set includes participants who had pre- and postvaccination blood samples within predefined day ranges, were seronegative to rubella at baseline, and followed protocol procedures.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 829 | 421 | 148
IU/mL | 98.7 [92.8 to 105.0] | 99.9 [91.8 to 108.7] | 126.3 [111.9 to 142.6]

14. Primary Outcome: Antibody Response to Varicella at 6 Weeks Postvaccination for Participants Initially Seronegative to Varicella at Baseline - GMT
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Varicella. (Titers measured using VZV gpELISA.)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 757 | 383 | 139
gpELISA units/mL | 13.8 [12.8 to 14.8] | 15.4 [13.8 to 17.0] | 15.8 [13.8 to 18.0]

15. Primary Outcome: Antibody Response to Diphtheria at 6 Weeks Postvaccination - GMT
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Diphtheria. (Titers measured using Vero Cell Culture Assay.)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 675 | 337 | 95
IU/mL | 1.33 [1.24 to 1.43] | 1.72 [1.55 to 1.89] | 1.59 [1.29 to 1.97]

16. Primary Outcome: Antibody Response to Pertussis Toxin (PT) at 6 Weeks Postvaccination - GMT
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Pertussis Toxin (PT). Titers measured using an indirect, noncompetitive Pertussis enzyme immunoassay (EIA).
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: units/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 748 | 355 | 59
units/mL | 42.9 [39.5 to 46.5] | 55.7 [49.7 to 62.4] | 46.3 [35.0 to 61.4]

17. Primary Outcome: Antibody Response to Pertussis Filamentous Hemagglutinin (FHA) at 6 Weeks Postvaccination - GMT
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Pertussis Filamentous Hemagglutinin (FHA). (Titers measured using an indirect, noncompetitive Pertussis enzyme immunoassay (EIA).)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: units/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 748 | 356 | 59
units/mL | 58.1 [53.7 to 62.9] | 81.2 [73.5 to 89.7] | 65.0 [49.6 to 85.2]

18. Primary Outcome: Antibody Response to Hepatitis B at 6 Weeks Postvaccination - GMT
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Hepatitis B. (Titers measured using the Quantitative AUSAB™ radioimmunoassay (RIA).)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 825 | 396 | 122
mIU/mL | 758 [658 to 874] | 996 [828 to 1199] | 1135 [836 to 1541]

19. Primary Outcome: Antibody Response to Haemophilus Influenzae Type B (Hib) at 6 Weeks Postvaccination - GMT
Description: Postvaccination observed GMT of antibody to Hib. (Anti-polyribosylribitol phosphate (PRP) was measured by RIA using radiolabeled-PRP according to a standard Farr technique and with a standard provided by the U.S. FDA.)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 822 | 398 | 124
mIU/mL | 11.2 [10.1 to 12.3] | 12.1 [10.6 to 13.7] | 12.9 [10.4 to 16.1]

20. Primary Outcome: Antibody Response to Tetanus at 6 Weeks Postvaccination - GMT
Description: Postvaccination Observed Geometric Mean Titer of Antibody to Tetanus. (Titers of tetanus antitoxin were measured with an indirect, noncompetitive enzyme immunoassay (EIA).)
Time Frame: 6 weeks Postvaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Number analyzed (Participants) | 803 | 387 | 114
IU/mL | 3.93 [3.59 to 4.31] | 5.74 [5.13 to 6.42] | 4.36 [3.67 to 5.17]

ADVERSE EVENTS:
Time Frame: Participants were followed for safety for 42 days after Visit 1 and 14 days after Visit 2 (56 days total).
Description: Number of participants reported as "At Risk" is the number of participants with follow-up.
  Although a subject may have had 2 or more adverse experiences, the subject is counted only once within a category. The same subject may appear in different categories.
Arm/Group | Concomitant Group | Nonconcomitant Group | Control Group
Serious Adverse Events (participants affected / at risk) | 11/929 | 3/479 | 1/467
Other Adverse Events (participants affected / at risk) | 831/929 | 435/479 | 411/467
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concomitant Group (N=929) | Nonconcomitant Group (N=479) | Control Group (N=467)
Fever (General disorders) | 0 | 1 | 0
Hernia, inguinal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Infection, viral (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Allergy, food (Immune system disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Afebrile seizure (Nervous system disorders) | 1 | 0 | 1
Seizure, febrile (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Laryngotracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cellulitis, orbital (Infections and infestations) | 1 | 0 | 0
Necrosis, testicle (Reproductive system and breast disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Concomitant Group (N=929) | Nonconcomitant Group (N=479) | Control Group (N=467)
Fever (General disorders) | 295 | 142 | 136
Infection, Viral (Infections and infestations) | 41 | 27 | 18
Malaise (General disorders) | 5 | 2 | 6
Pain (General disorders) | 11 | 2 | 4
Trauma (Injury, poisoning and procedural complications) | 13 | 3 | 6
Anorexia (Metabolism and nutrition disorders) | 17 | 12 | 5
Constipation (Gastrointestinal disorders) | 3 | 4 | 5
Diarrhea (Gastrointestinal disorders) | 88 | 33 | 48
Flatulence (Gastrointestinal disorders) | 12 | 4 | 5
Gastroenteritis (Gastrointestinal disorders) | 18 | 4 | 9
Gastroenteritis, Infectious (Infections and infestations) | 17 | 5 | 7
Vomiting (Gastrointestinal disorders) | 56 | 31 | 30
Allergy (Immune system disorders) | 9 | 4 | 6
Irritability (Psychiatric disorders) | 109 | 52 | 67
Asthma (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 5
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 7
Congestion, Nasal (Respiratory, thoracic and mediastinal disorders) | 16 | 16 | 9
Congestion, Respiratory (Respiratory, thoracic and mediastinal disorders) | 29 | 13 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 83 | 47 | 43
Infection, Respiratory, Upper (Infections and infestations) | 258 | 131 | 108
Influenza (Infections and infestations) | 5 | 3 | 7
Laryngotracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 24 | 11 | 6
Rhinitis (Reproductive system and breast disorders) | 16 | 14 | 10
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 64 | 32 | 41
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 19 | 8 | 17
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11 | 5 | 6
Bite/Sting, Non-Venomous (Injury, poisoning and procedural complications) | 20 | 12 | 10
Contusion (Injury, poisoning and procedural complications) | 5 | 6 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 8 | 1 | 6
Dermatitis, Contact (Skin and subcutaneous tissue disorders) | 11 | 10 | 4
Eczema (Skin and subcutaneous tissue disorders) | 16 | 7 | 8
Excoriation (Skin and subcutaneous tissue disorders) | 1 | 2 | 5
Miliaria Rubra (Skin and subcutaneous tissue disorders) | 44 | 16 | 17
Rash (Skin and subcutaneous tissue disorders) | 45 | 22 | 25
Rash, Diaper (Skin and subcutaneous tissue disorders) | 82 | 37 | 43
Rash, Measles/Rubella-Like (Skin and subcutaneous tissue disorders) | 27 | 16 | 10
Rash, Varicella-Like (Skin and subcutaneous tissue disorders) | 13 | 12 | 15
Urticaria (Skin and subcutaneous tissue disorders) | 13 | 4 | 6
Viral Exanthema (Infections and infestations) | 71 | 25 | 23
Conjunctivitis (Eye disorders) | 27 | 21 | 18
Otitis (Ear and labyrinth disorders) | 60 | 19 | 13
Otitis Media (Ear and labyrinth disorders) | 175 | 83 | 77
Pain, Ear (Ear and labyrinth disorders) | 4 | 3 | 5
Ecchymosis (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 17 | 10 | 0/0
Erythema (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 165 | 83 | 0/0
Pain/Tenderness/Soreness (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 308 | 121 | 0/0
Rash (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 11 | 9 | 0/0
Swelling (ProQuad Injection-site) (Skin and subcutaneous tissue disorders) | 115 | 51 | 0/0
Erythema (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 56
Pain/Tenderness/Soreness (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 121
Swelling (Varivax Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 28
Erythema (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 64
Pain/Tenderness/Soreness (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 125
Swelling (M-M-R II Injection-site) (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 32
Ecchymosis (Tripedia Injection-site) (Skin and subcutaneous tissue disorders) | 10 | 7 | 3
Erythema (Tripedia Injection-site) (Skin and subcutaneous tissue disorders) | 244 | 113 | 110
Pain/Tenderness/Soreness (Tripedia Injection-site) (Skin and subcutaneous tissue disorders) | 327 | 134 | 140
Swelling (Tripedia Injection-site) (Skin and subcutaneous tissue disorders) | 203 | 83 | 78
Ecchymosis (Comvax Injection-site) (Skin and subcutaneous tissue disorders) | 11 | 4 | 1
Erythema (Comvax Injection-site) (Skin and subcutaneous tissue disorders) | 266 | 118 | 113
Induration (Comvax Injection-site) (Skin and subcutaneous tissue disorders) | 8 | 2 | 7
Pain/Tenderness/Soreness (Comvax Injection-site) (Skin and subcutaneous tissue disorders) | 327 | 143 | 139
Swelling (Comvax Injection-site) (Skin and subcutaneous tissue disorders) | 204 | 84 | 82

LIMITATIONS AND CAVEATS:
Two participants were incorrectly vaccinated and are not included in the efficacy/safety analyses. One received M-M-R™II+TRIPEDIA™+COMVAX™ and 1 received VARIVAX™+TRIPEDIA™+COMVAX™ instead of ProQuad™+TRIPEDIA™+COMVAX™

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.